CLINICAL TRIAL: NCT06995261
Title: The Performance of an Individual Dosing Regimen of Follitropin Delta (Fd) in a GnRH Agonist Protocol for Controlled Ovarian Stimulation for IVF/ICSI in a Real-word Setting: a Non-interventional Cohort Study
Brief Title: Follitropin Delta in Long GnRH-agonist Protocol
Acronym: REWAG
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. med. M.Sc. Georg Griesinger (Other)
Collaborators: University Hopsital Schleswig Holstein Campus Lübeck (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. M.Sc. Georg Griesinger, Professor of Gynecological Endocrinology and Reproductive Medicine, Director, IVF Center, University of Lübeck / UKSH, University of Luebeck
Organization: University of Luebeck (Other)
Other Study IDs: 2025-123 EC Luebeck
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Infertility (IVF Patients); Infertility; Infertility Drugs
Keywords: follitropin delta; Rekovelle; Long GnRH-agonist protocol; individualized ovarian stimulation; Dosing algorithm; FSH
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follitropin Delta in Long GnRH Agonist Protocol: This cohort includes women undergoing controlled ovarian stimulation for IVF or ICSI treatment using Follitropin delta administered in a long GnRH agonist protocol. The dosing is individualized based on AMH serum levels and body weight. Participants are treated according to routine clinical practice, and no study drug is provided. The study is non-interventional.

SUMMARY:
The REWAG study ("Real-world Evaluation of Women undergoing Agonist protocol with Follitropin delta") is a non-interventional observational study conducted across several fertility centers in Germany. The goal of this study is to evaluate how well a personalized dosing regimen of a hormone called Follitropin delta works in women undergoing controlled ovarian stimulation (COS) for in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) using a long GnRH agonist protocol.

Follitropin delta is a recombinant follicle-stimulating hormone (rFSH) that allows for individualized dosing based on a woman's weight and a blood marker called anti-Müllerian hormone (AMH). This personalized approach may help to better balance the stimulation of the ovaries, aiming to reduce the risk of overstimulation (OHSS) while still achieving good treatment outcomes.

The study will include approximately 350 women who are undergoing routine IVF/ICSI treatment. No experimental drugs or procedures are involved. All treatment decisions remain the responsibility of the attending physicians and follow standard clinical practice. Data will be collected only from routine visits and medical documentation, with no additional interventions required for participation.

Researchers will analyze outcomes such as the number of eggs retrieved, pregnancy rates, treatment cancellations, and any side effects. The study will also look at whether certain patient characteristics can predict how well the treatment works or whether complications may arise.

Participation is voluntary. All personal data will be pseudonymized and handled according to strict data protection regulations (GDPR). Results will help to improve understanding of how personalized hormone dosing performs in real-life settings and may support more tailored and effective fertility treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to ≤ 44 years at enrolment
* Planned stimulation in a long luteal GnRH agonist protocol with daily s.c. GnRH-agonist
* Planned use of Fd for ovarian stimulation as per SmPC
* Serum AMH ≥0.3 ng/ml to ≤4.9 ng/ml measured within12 months prior to treatment
* Most recent serum AMH value before start of stimulation not older than 12 months
* Planned IVF or ICSI treatment in a first or second attempt with ejaculated or cryopreserved male germ cells, autologous or heterologous, with or without planned genetic testing of the oocytes or embryos
* Planned triggering of final oocyte maturation with hCG
* Willingness and consent to participate

Exclusion Criteria:

* Serum AMH value not determined in ELECSYS AMH Plus Immunoassay, ACCESS AMH Advanced (Beckham Coulter) or LUMIPULSE G AMH (Fujirebio)
* Most recent serum AMH value before start of stimulation older than 12 months
* Serum AMH within 12 months prior to treatment AMH ≤ 0.3 ng/ml or ≥4.9 ng/ml measured within 12 months prior to treatment
* Pre-treatment with a combined oral contraceptive "pill" consisting of ethinyl estradiol and a synthetic progestogen or a natural estradiol/progesterone
* Anovulatory PCOS syndrome
* Women with a contraindication for prescription of Fd treatment
* Women undergoing ovarian stimulation for fertility preservation

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women undergoing IVF oder ICSI. This study is intended to be conducted in non-vulnerable population. No vulnerable subjects will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Ovarian Hyperstimulation Syndrome (OHSS) | From oocyte pick-up to gestational week 20
  Ovarian Hyperstimulation Syndrome (OHSS) of any grade and any onset by Golan classification

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Department of Obstetrics, Gynecology and Reproductive Endocrinology (UniKiD), Medical Faculty and University Hospital Düsseldorf, Heinrich Heine University Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Center for Reproductive Medicine, IVF SAAR, Saarbrücken, Saarland
  - Department of Reproductive Medicine and Gynecological Endocrinology, University Hospital of Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Department of Reproductive Medicine and Gynecological Endocrinology, University Hospital of Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lobo R, Soerdal T, Ekerhovd E, Cohlen B, Porcu E, Schenk M, Shufaro Y, Smeenk J, Suerdieck MB, Pinton P, Pinborg A; BEYOND Investigators. BEYOND: a randomized controlled trial comparing efficacy and safety of individualized follitropin delta dosing in a GnRH agonist versus antagonist protocol during the first ovarian stimulation cycle. Hum Reprod. 2024 May 9;39(7):1481-94. doi: 10.1093/humrep/deae092. Online ahead of print. PMID 38723189